CLINICAL TRIAL: NCT04012697
Title: A Randomized Controlled Trial of Peer Support Workers in the Emergency Department for People Experiencing Homelessness in the Niagara Region of Ontario, Canada
Brief Title: Peer Support for Homelessness in the Emergency Department
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: McMaster University (Other)
Collaborators: Niagara Community Foundation (Unknown); United Way Niagara (Unknown); Niagara Poverty Reduction Network (Unknown); Quest Community Health Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 7048
Record Dates: First submitted 2019-07-02; First posted 2019-07-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Homelessness; Health Behavior; Health Care Utilization; Health Care Seeking Behavior
Keywords: Survival analysis; Quantitative analysis; Patient-reported outcomes; Randomized-controlled trial; Homelessness; Health services research; Administrative health data; Peer support
MeSH Terms: conditions — Health Behavior; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized controlled superiority trial with parallel intervention and usual care groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Baseline data collection is performed prior to randomization and group assignment. Data collection at each of the following Time points is performed by research assistants who are blinded to the participant's group assignment. Investigators are likewise blinded to the group assignment of participants. Participants are not blinded given the impracticality of blinding assignment to the group receiving peer support vs. receiving usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Support (Experimental): Peer support services from a peer support worker in the emergency department.
  Interventions: Behavioral: Peer Support
- Usual care (No Intervention): Usual care in the emergency department.

INTERVENTIONS:
Behavioral: Peer Support — Participants randomized to the intervention group will be seen by the peer support worker during their stay in the emergency department. The goal of the peer support worker's practice is to address the participant's wellness from a holistic point of view that includes their relationships, connections to the community, general well-being, and sense of empowerment, with an overall focus on quality-of-life goals (Sunderland et al., 2013). The peer support worker will provide a multi-faceted intervention, which aims to foster a peer-to-peer relationship encompassing elements of empathic communication, brief supportive counseling, advocacy for non-medical needs in hospital, liaising and collaborating with medical and nursing staff, motivational interviewing, and connection with programs in the community.
  Arms: Peer Support

SUMMARY:
Peer support workers with lived experience of homelessness will provide advocacy, supportive counselling, assistance with navigating the system, and role-modeling for people experiencing homelessness in emergency departments in the Niagara region of Ontario, Canada. Previous research has demonstrated that people experiencing homelessness experience barriers to care and poor health outcomes, including increased risk of dying, and are frequent users of the emergency department for physical and mental health needs. The benefits of peer support have been studied in hospital psychiatric units and with people experiencing homelessness, but no studies have yet explored the potential impact of peer support workers on homelessness in the emergency department. The investigators plan to do a 12-month randomized study of peer support workers compared to usual care in the emergency department, and evaluate outcomes such as physical health, mental health, addictions, and behaviours, as well as cost-effectiveness and changes in how people experiencing homelessness seek health care. The investigators hope that the findings of this study will provide additional knowledge and evidence for future efforts to improve care for people experiencing homelessness.

DETAILED DESCRIPTION:
Homelessness is strongly associated with an increased prevalence of chronic physical and mental health morbidity, leading to lower health-related quality of life and increased hospital readmissions compared to the general population. People experiencing homelessness have reported experience of discrimination and unwelcome treatment, neglect and rejection, lack of compassion from their health care providers and feeling as though their perceptions are disregarded. Alongside many daily barriers such as substance use, lack of housing, and food insecurity, these issues also negatively influence the desire to seek health care among people experiencing homelessness.

A national strategy to determine the extent and nature of homelessness, 'Point-in-Time Counts' were conducted in over 60 communities across Canada in 2018 to provide a snapshot of the experiences and needs of people experiencing homelessness. The Niagara 'Point-in-Time' Count collected 408 surveys from people experiencing homelessness, with 57 percent of participants reporting a mental health issue, 36.2 percent reporting an addiction, and 33.9 percent reporting a medical condition. Respondents also reported an ongoing need for mental health services (54.3 percent), addiction services (29.2 percent), and medical services (26.9 percent). Of note, 219 participants reporting a collective 663 visits to the emergency department in the preceding 12 months. People experiencing homelessness are much more likely than housed people to access emergency departments for concerns with mental health, although this may not be an ideal environment to provide recovery-based mental health care.

The placement of peer support workers in the emergency department may help overcome barriers to health care for people experiencing homelessness. Peer support is defined as a supportive relationship between a worker and a peer who share the commonality of a lived experience, with the peer support worker able to model recovery and use a recovery-oriented, person-centered approach with their peer. Increasing positive interactions in a clinical care setting could address the lack of trust perceived by people experiencing homelessness towards health care providers, helping to counteract negative perceptions of health care and increasing the likelihood that people experiencing homelessness will seek care in the future.

The benefits of a peer support worker include feelings of empowerment and hope, increased sense of acceptance and empathy, improved satisfaction, and reduced feelings of stigma. Peer support workers in mental health services lead to reduced admissions, as well as earlier discharge when utilized following admission to hospital. Two recent reviews investigated the effectiveness of peer support services in individuals with severe mental illness. Consistently, they found that peers are at least as effective in providing services as non-peers in the same roles. Additionally, there are certain unique elements that can only be provided by peer support workers. Three randomized controlled trials reported better treatment engagement, fewer hospitalizations and hospital days, and lower rates of non-attendance compared to treatment as usual when peer support workers were added to a care team. When peer support workers served as patient advocates and community connectors for people with multiple psychiatric hospitalizations, the number of hospitalizations and days spent in hospital decreased. Furthermore, participants reported a decrease in depressive symptoms and increase in hope, self-care, and sense of well-being. The researchers noted that the active ingredient in these interventions seemed to be the instillation of hope through self-disclosure, role modeling, and empathy paired with conditional regard. Upon comparing and contrasting the core competencies of case managers and peer support workers, it was noted that the unique duties of peer support workers seemed to center around empowering clients via normalization, participating in personal development as a role model, and encouraging clients' educational growth.

However, despite promising findings in a diversity of clinical care settings, there has been relatively limited research and few high quality studies of the effectiveness of peer support workers and their outcomes with people experiencing homelessness. People experiencing homelessness typically have complex comorbid mental illnesses, and they should theoretically benefit from peer support services via the sharing of lived experiences. An exploratory review of the literature on peer support and homelessness found 10 studies totaling 1341 participants that collectively reported improved overall quality of life, significant increases in social support, reduced rates of substance use, decreased homelessness, and better physical and mental health for the recipients of peer support. Although promising, six of the included studies were longitudinal, two were cross-sectional, and two were quasi-experimental. There was also significant heterogeneity in the delivery of peer services across studies, including peer support from mentors, peer support as part of a larger intervention, and peer support groups.

Within the emergency department, there has been minimal research on peer support or similar interventions. Of 11 studies examined in a meta-analysis of the effectiveness of emergency department interventions for frequent users, case management was found to be the most frequently used. For people experiencing homelessness, case management demonstrated increased contact with health services, reduced lengths of admission, decreased emergency department visits for mental health problems, and reduced substance use, but only equivocal findings for physical and mental health. An example of an emergency department program that is similar to peer support can be found in a randomized trial of compassionate care for people experiencing homelessness. This study from 1995 found that compassionate contact from trained volunteers led to a 33% relative reduction in the overall frequency of visits per month and a significant reduction in the time until a first repeat visit; however, health outcomes were not evaluated.

Although there are several types of emergency department interventions, there is overall a lack of evidence about program effectiveness. Very few studies are randomized controlled trials, most studies with high-risk individuals are of low quality, and stronger evidence on cost-effectiveness is necessary for all program types. Furthermore, the quality of care and health outcomes for people experiencing homelessness may be improved through peer support, but evidence in this area is underdeveloped and in need of studies with robust experimental measures. To fill this gap in knowledge, this study will evaluate a program of peer support for people experiencing homelessness who seek care in the emergency departments of a mid-sized Canadian regional municipality. The research questions for the study are as follows:

1. What, if any, are the changes in health service use (e.g., emergency department visits, hospitalizations) following receipt of peer support in the emergency department?
2. What, if any, are the changes to health status, health-related quality of life, substance use, or behaviours, following engagement with a peer support worker?
3. Is peer support in the emergency department a cost-effective intervention?
4. Does receiving peer support in the emergency department lengthen the interval of time before a clinically significant outcome such as a repeat visit to the emergency department or increased morbidity?
5. What are the mechanisms of peer support in the emergency department that may contribute to differences observed in the outcomes between the intervention and usual care groups?

ELIGIBILITY:
Inclusion Criteria:

* Canadian citizen or permanent resident
* Resident of Ontario in the past 12 months
* Age 18 or over
* Absolute homeless (e.g., living outside, including but not limited to abandoned buildings, vehicles, transit stations; residing in shelters; residing in hotel/motel rooms)
* Hidden homeless (e.g., living with others, residing in transitional housing)

Exclusion Criteria:

* Not a Canadian citizen or permanent resident of Canada
* Not a resident of Ontario for the majority of the past 12 months
* Under the age of 18
* Does not meet criteria for absolute or hidden homelessness (see: Inclusion Criteria)
* Refusal to disclose housing, citizenship, or residential status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Change in mean from the pre-intervention 12-month baseline to the post-intervention 12-month period in the number of hospitalizations, measured using administrative health data | 12 months pre-study enrollment and 12-months post-study enrollment
  The primary outcome of the study includes the number of hospitalizations. This outcome will be evaluated through linkage and evaluation of administrative data hosted at Niagara Health through Decision Support Services. Consent will be obtained from participants to perform data linkage with Niagara Health databases and collect information on health services use for the 12-month period preceding and 12-month period following study enrollment.
Change in mean from the pre-intervention 12-month baseline to the post-intervention 12-month period in the number of days spent in hospital, measured using administrative health data | 12 months pre-study enrollment and 12-months post-study enrollment
  The primary outcome of the study includes the number of days spent in hospital. This outcome will be evaluated through linkage and evaluation of administrative data hosted at Niagara Health through Decision Support Services. Consent will be obtained from participants to perform data linkage with Niagara Health databases and collect information on health services use for the 12-month period preceding and 12-month period following study enrollment.
Change in mean from the pre-intervention 12-month baseline to the post-intervention 12-month period in the number of emergency department visits, measured using administrative health data | 12 months pre-study enrollment and 12-months post-study enrollment
  The primary outcome of the study includes the number of emergency department visits. This outcome will be evaluated through linkage and evaluation of administrative data hosted at Niagara Health through Decision Support Services. Consent will be obtained from participants to perform data linkage with Niagara Health databases and collect information on health services use for the 12-month period preceding and 12-month period following study enrollment.
Change in mean from the pre-intervention 12-month baseline to the post-intervention 12-month period in the number of hours spent in the emergency department at each visit, measured using administrative health data | 12 months pre-study enrollment and 12-months post-study enrollment
  The primary outcome of the study includes the number of hours spent in the emergency department at each visit. This outcome will be evaluated through linkage and evaluation of administrative data hosted at Niagara Health through Decision Support Services. Consent will be obtained from participants to perform data linkage with Niagara Health databases and collect information on health services use for the 12-month period preceding and 12-month period following study enrollment.
Change in mean from the pre-intervention 12-month baseline to the post-intervention 12-month period in the number of procedures performed in the emergency department, measured using administrative health data | 12 months pre-study enrollment and 12-months post-study enrollment
  The primary outcome of the study includes the number of procedures performed in the emergency department. This outcome will be evaluated through linkage and evaluation of administrative data hosted at Niagara Health through Decision Support Services. Consent will be obtained from participants to perform data linkage with Niagara Health databases and collect information on health services use for the 12-month period preceding and 12-month period following study enrollment.
Change in mean from the pre-intervention 12-month baseline to the post-intervention 12-month period in procedures performed during hospitalizations, measured using administrative health data | 12 months pre-study enrollment and 12-months post-study enrollment
  The primary outcome of the study includes the number of procedures performed during hospitalizations. This outcome will be evaluated through linkage and evaluation of administrative data hosted at Niagara Health through Decision Support Services. Consent will be obtained from participants to perform data linkage with Niagara Health databases and collect information on health services use for the 12-month period preceding and 12-month period following study enrollment.
Change in proportions from the pre-intervention 12-month baseline to the post-intervention 12-month period in diagnoses at the time of discharge from the emergency department, measured using administrative health data | 12 months pre-study enrollment and 12-months post-study enrollment
  The primary outcome of the study includes the diagnosis at time of discharge from the emergency department. This outcome will be evaluated through linkage and evaluation of administrative data hosted at Niagara Health through Decision Support Services. Consent will be obtained from participants to perform data linkage with Niagara Health databases and collect information on health services use for the 12-month period preceding and 12-month period following study enrollment.
Change in proportion from the pre-intervention 12-month baseline to the post-intervention 12-month period in mortality, measured using administrative health data | 12 months pre-study enrollment and 12-months post-study enrollment
  The primary outcome of the study includes mortality. This outcome will be evaluated through linkage and evaluation of administrative data hosted at Niagara Health through Decision Support Services. Consent will be obtained from participants to perform data linkage with Niagara Health databases and collect information on health services use for the 12-month period preceding and 12-month period following study enrollment.
Change in proportion from the pre-intervention 12-month baseline to the post-intervention 12-month period in overdose presentations, measured using administrative health data | 12 months pre-study enrollment and 12-months post-study enrollment
  The primary outcome of the study includes overdose presentations. This outcome will be evaluated through linkage and evaluation of administrative data hosted at Niagara Health through Decision Support Services. Consent will be obtained from participants to perform data linkage with Niagara Health databases and collect information on health services use for the 12-month period preceding and 12-month period following study enrollment.
Change in proportion from the pre-intervention 12-month baseline to the post-intervention 12-month period in psychiatric presentations, measured using administrative health data | 12 months pre-study enrollment and 12-months post-study enrollment
  The primary outcome of the study includes psychiatric presentations. This outcome will be evaluated through linkage and evaluation of administrative data hosted at Niagara Health through Decision Support Services. Consent will be obtained from participants to perform data linkage with Niagara Health databases and collect information on health services use for the 12-month period preceding and 12-month period following study enrollment.
Change in proportion from pre-intervention 12-month baseline to post-intervention 12-month period in composition of presenting complaints to the emergency department, measured using administrative health dat | 12 months pre-study enrollment and 12-months post-study enrollment
  The primary outcome of the study includes the composition of presenting complaints to the emergency department and potential differences over time in the proportions of different presentations (e.g., physical health vs. mental health, Canadian Triage and Acuity Scale (CTAS) levels). This outcome will be evaluated through linkage and evaluation of administrative data hosted at Niagara Health through Decision Support Services. Consent will be obtained from participants to perform data linkage with Niagara Health databases and collect information on health services use for the 12-month period preceding and 12-month period following study enrollment.

SECONDARY OUTCOMES:
Mean change from baseline in psychiatric symptoms on the Colorado Symptom Index (CSI) at 6 months | 6 months
  The CSI is a 14-item self-report measure of psychiatric symptoms (Boothroyd & Chen, 2008). Respondents report the frequency of various psychiatric symptoms as experienced over the past month on a 5-point Likert scale. Scores range from 0 to 56, with higher scores indicating report of more frequent psychiatric symptoms. The CSI has been psychometrically validated with a sample of people who were experiencing homelessness, living precariously, at risk for homelessness, or had prior history of homelessness (Conrad et al., 2001). The CSI was found to have excellent internal consistency with a Cronbach's alpha of 0.90 and a test/retest intraclass correlation coefficient of 0.79 with this population. The CSI is intended to evaluate change in persons with moderate and high severity psychological symptoms or emotional distress, and is sensitive to change in symptomatology over time. Administration of the questionnaire requires approximately 5 minutes.
Mean change from baseline in psychiatric symptoms on the Colorado Symptom Index (CSI) at 12 months | 12 months
  The CSI is a 14-item self-report measure of psychiatric symptoms (Boothroyd & Chen, 2008). Respondents report the frequency of various psychiatric symptoms as experienced over the past month on a 5-point Likert scale. Scores range from 0 to 56, with higher scores indicating report of more frequent psychiatric symptoms. The CSI has been psychometrically validated with a sample of people who were experiencing homelessness, living precariously, at risk for homelessness, or had prior history of homelessness (Conrad et al., 2001). The CSI was found to have excellent internal consistency with a Cronbach's alpha of 0.90 and a test/retest intraclass correlation coefficient of 0.79 with this population. The CSI is intended to evaluate change in persons with moderate and high severity psychological symptoms or emotional distress, and is sensitive to change in symptomatology over time. Administration of the questionnaire requires approximately 5 minutes.
Mean change from baseline in psychopathology and crime/violence on the Global Appraisal of Individual Needs - Short Screener (GAIN-SS) at 6 months | 6 months
  The GAIN-SS is a 24-item self-report measure which assesses psychopathology and crime/violence across various dimensions and screens for people who are likely to have diagnoses or require clinical services (Dennis, Chan, & Funk, 2006). The total score contributes to a Total Disorder Screener (TDScr), with four, 5- to 7-item subset screeners including the Internalizing Disorder Screener (IDScr), Externalizing Disorder Screener (EDScr), Substance Disorder Screener (SDScr), and Crime/Violence Screener (CVScr). The GAIN-SS is internally consistent with a Cronbach's alpha of 0.89 and good discriminant validity for each of the sub-screeners. The Total Disorder Screener has over 90% sensitivity and specificity with a ROC of 0.97 with a cut point of 3 or more. For the sub-screeners, scores can be divided into three groupings of 0 (low), 1-2 (moderate), and 3-5 (high), with the lower cut point of 1+ featuring 90% sensitivity and the upper cut point of 3+ featuring 90% specificity.
Mean change from baseline in psychopathology and crime/violence on the Global Appraisal of Individual Needs - Short Screener (GAIN-SS) at 12 months | 12 months
  The GAIN-SS is a 24-item self-report measure which assesses psychopathology and crime/violence across various dimensions and screens for people who are likely to have diagnoses or require clinical services (Dennis, Chan, & Funk, 2006). The total score contributes to a Total Disorder Screener (TDScr), with four, 5- to 7-item subset screeners including the Internalizing Disorder Screener (IDScr), Externalizing Disorder Screener (EDScr), Substance Disorder Screener (SDScr), and Crime/Violence Screener (CVScr). The GAIN-SS is internally consistent with a Cronbach's alpha of 0.89 and good discriminant validity for each of the sub-screeners. The Total Disorder Screener has over 90% sensitivity and specificity with a ROC of 0.97 with a cut point of 3 or more. For the sub-screeners, scores can be divided into three groupings of 0 (low), 1-2 (moderate), and 3-5 (high), with the lower cut point of 1+ featuring 90% sensitivity and the upper cut point of 3+ featuring 90% specificity.
Mean change from baseline in health status on the EuroQol-5D-5L (EQ-5D-5L) at 6 months | 6 months
  The EQ-5D is a 5-item generic measure of health status that provides a descriptive profile for respondents to provide a self-rating of their health and produce a utility score for cost-effectiveness analysis. Health is defined across five dimensions of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, which encompass a broad range of different disease areas, specialties, and types of care. Each dimension offers the following five levels: No problems, slight problems, moderate problems, severe problems, and unable to/extreme problems. The EQ-5D-5L offers a total of 3125 health states with a value set for Canada demonstrating a range of health utilities from -0.148 for the worst health state (55555, that is, extreme problems with mobility, self-care, etc.) to 0.949 for the best health state (11111, that is, no problems with any of the dimensions).
Mean change from baseline in health status on the Visual Analogue Scale (VAS) at 6 months | 6 months
  The Visual Analogue Scale is a 20-cm scale for respondents to provide a self-rating of their health and produce a utility score for cost-effectiveness analysis. This instrument offers a total of 3125 health states with a value set for Canada demonstrating a range of health utilities from -0.148 for the worst health state (55555, that is, extreme problems with mobility, self-care, etc.) to 0.949 for the best health state (11111, that is, no problems with any of the dimensions).
Mean change from baseline in health status on the EuroQol-5D-5L (EQ-5D-5L) at 12 months | 12 months
  The EQ-5D is a 5-item generic measure of health status that provides a descriptive profile for respondents to provide a self-rating of their health and produce a utility score for cost-effectiveness analysis. Health is defined across five dimensions of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, which encompass a broad range of different disease areas, specialties, and types of care. Each dimension offers the following five levels: No problems, slight problems, moderate problems, severe problems, and unable to/extreme problems. The EQ-5D-5L offers a total of 3125 health states with a value set for Canada demonstrating a range of health utilities from -0.148 for the worst health state (55555, that is, extreme problems with mobility, self-care, etc.) to 0.949 for the best health state (11111, that is, no problems with any of the dimensions).
Mean change from baseline in health status on the Visual Analogue Scale (VAS) at 12 months | 12 months
  The Visual Analogue Scale is a 20-cm scale for respondents to provide a self-rating of their health and produce a utility score for cost-effectiveness analysis. This instrument offers a total of 3125 health states with a value set for Canada demonstrating a range of health utilities from -0.148 for the worst health state (55555, that is, extreme problems with mobility, self-care, etc.) to 0.949 for the best health state (11111, that is, no problems with any of the dimensions).
Mean change from baseline in mental health and physical health on the 12-item Short Form Survey (SF-12) at 6 months | 6 months
  The SF-12 is a 12-item questionnaire that has been investigated and utilized for measuring health status among people experiencing homelessness (Larson, 2002). It features categorical questions that assess limitations in role functioning as a result of physical and emotional health, as well as numerous Likert scale responses including a 3-point scale to assess limitations in physical activity and physical role functioning, a 5-point scale for pain and another for overall health, and a 6-point scale to assess mental health, vitality, and social functioning. The SF-12 produces a summary score each for mental health and physical health, which are able to differentiate between diagnostic groups and levels of severity of illness. Internal consistency in a sample of people experiencing homelessness demonstrated a Cronbach's alpha of 0.82 for physical health and 0.79 for mental health.
Mean change from baseline in mental health and physical health on the 12-item Short Form Survey (SF-12) at 12 months | 12 months
  The SF-12 is a 12-item questionnaire that has been investigated and utilized for measuring health status among people experiencing homelessness (Larson, 2002). It features categorical questions that assess limitations in role functioning as a result of physical and emotional health, as well as numerous Likert scale responses including a 3-point scale to assess limitations in physical activity and physical role functioning, a 5-point scale for pain and another for overall health, and a 6-point scale to assess mental health, vitality, and social functioning. The SF-12 produces a summary score each for mental health and physical health, which are able to differentiate between diagnostic groups and levels of severity of illness. Internal consistency in a sample of people experiencing homelessness demonstrated a Cronbach's alpha of 0.82 for physical health and 0.79 for mental health.

OTHER OUTCOMES:
Cost-effectiveness analysis of peer support worker intervention as compared to usual care at 12 months | 12 months
  The total mean costs for the usual care group will be subtracted from the total mean costs for the intervention group to provide the incremental cost (IC). The mean quality-adjusted life years (QALYs) associated with the intervention and usual care groups will be calculated using the health state and associated health utility score from the Time 12 administration of the EQ-5D-5L, multiplied against the value of '1' representing a 12-month treatment effect/duration of peer support (or usual care). The mean QALY of the usual care group will be subtracted from the mean QALY of the intervention group to provide the incremental effectiveness (IE). The incremental cost-effectiveness ratio (ICER), representing the average cost per additional QALY gained, will be calculated by dividing IC by IE (Neumann, Sanders, Russell, Siegel, & Ganiats, 2017).
Survival analysis of health service use/outcomes using administrative health data | From the date of assignment until the date of first emergency department readmit, second emergency department readmit, and admission to an inpatient service, assessed up to 12 months
  We will examine time to first emergency department readmit, time to second emergency department readmit, and time to admission to an inpatient service. A failure is considered to have occurred if the participant visits the emergency department after the enrollment presentation or is admitted to hospital through the emergency department.
Non-parametric survival analysis using administrative health and peer support questionnaire data to evaluate changes in health care provision between contacts with the peer support worker | From the date of assignment until the date of each subsequent visit, assessed up to 12 months
  We will examine the amount of procedures, tests and time spent within an emergency department as a crude measurement of health needs. At first presentation, an increase in these values in the intervention group relative to the usual care group is suggestive that the peer support worker is providing information to the medical team that improves care. At subsequent visits though, if our intervention is effective at improving un-met health needs, the opposite relationship should occur. We will augment these administrative measures with aspects of an 11-item peer support worker survey which will further document interactions with the medical team.
Survival analysis of mental health and physical health on the SF-12 | From the date of assignment until the date of scoring one standard deviation below mean and two standard deviations below mean for each of physical health score and mental health score, respectively, assessed up to 12 months
  Survival analysis will be also conducted on the SF-12 to evaluate how quickly mental and physical health degrades in our sample after the initial intervention. We will count an occurrence of one and two standard deviations below mean as a failure in our sample and will perform this analysis on both physical and mental well-being summary scores separately.
Non-parametric survival analysis using data on address of residence to evaluate changes in discharge planning between contacts with the peer support worker | From the date of assignment until the date of address change designating a stay at a shelter or address change from previous contact, assessed up to 12 months
  We will assess discharge planning as a cause for improved health care system use. One reflection of improved discharge planning may be stability in the participant's address. Our strategy for data collection will include a question on the participant's address, and any other changes in their contact information. We will employ non-parametric survival analysis to see if our intervention is 1) Associated with reduced stays at shelters, and 2) Associated with the same address as previous contact. An outcome is considered a failure if the person is staying at a shelter or has changed addresses from previous contact.

CONTACTS AND LOCATIONS:
Overall Officials: Suneel Upadhye, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Academy of Peer Services. (n.d.). Retrieved December 23, 2018, from https://www.academyofpeerservices.org/
- [Background] Acosta O, Toro PA. Let's ask the homeless people themselves: a needs assessment based on a probability sample of adults. Am J Community Psychol. 2000 Jun;28(3):343-66. doi: 10.1023/A:1005105421548. PMID 10945121
- [Background] Althaus F, Paroz S, Hugli O, Ghali WA, Daeppen JB, Peytremann-Bridevaux I, Bodenmann P. Effectiveness of interventions targeting frequent users of emergency departments: a systematic review. Ann Emerg Med. 2011 Jul;58(1):41-52.e42. doi: 10.1016/j.annemergmed.2011.03.007. PMID 21689565
- [Background] Amato S, Nobay F, Amato DP, Abar B, Adler D. Sick and unsheltered: Homelessness as a major risk factor for emergency care utilization. Am J Emerg Med. 2019 Mar;37(3):415-420. doi: 10.1016/j.ajem.2018.06.001. Epub 2018 Jun 2. PMID 29891125
- [Background] Barker SL, Maguire N. Experts by Experience: Peer Support and its Use with the Homeless. Community Ment Health J. 2017 Jul;53(5):598-612. doi: 10.1007/s10597-017-0102-2. Epub 2017 Feb 7. PMID 28176210
- [Background] Boothroyd RA, Chen HJ. The psychometric properties of the Colorado Symptom Index. Adm Policy Ment Health. 2008 Sep;35(5):370-8. doi: 10.1007/s10488-008-0179-6. Epub 2008 Jun 17. PMID 18561020
- [Background] Broglio K. Randomization in Clinical Trials: Permuted Blocks and Stratification. JAMA. 2018 Jun 5;319(21):2223-2224. doi: 10.1001/jama.2018.6360. No abstract available. PMID 29872845
- [Background] Bungay V. Health care among street-involved women: the perpetuation of health inequity. Qual Health Res. 2013 Aug;23(8):1016-26. doi: 10.1177/1049732313493352. Epub 2013 Jun 12. PMID 23761930
- [Background] Cameron, A & Trivedi, P. (2005). Microeconometrics: Methods and applications. Cambridge: Cambridge University Press. Retrieved from https://ebookcentral.proquest.com.
- [Background] Conrad KJ, Yagelka JR, Matters MD, Rich AR, Williams V, Buchanan M. Reliability and validity of a modified Colorado Symptom Index in a national homeless sample. Ment Health Serv Res. 2001 Sep;3(3):141-53. doi: 10.1023/a:1011571531303. PMID 11718206
- [Background] Cook JA, Julious SA, Sones W, Hampson LV, Hewitt C, Berlin JA, Ashby D, Emsley R, Fergusson DA, Walters SJ, Wilson ECF, Maclennan G, Stallard N, Rothwell JC, Bland M, Brown L, Ramsay CR, Cook A, Armstrong D, Altman D, Vale LD. DELTA2 guidance on choosing the target difference and undertaking and reporting the sample size calculation for a randomised controlled trial. Trials. 2018 Nov 5;19(1):606. doi: 10.1186/s13063-018-2884-0. PMID 30400926
- [Background] Cousins, C. (2018). Niagara Counts. Retrieved from Niagara Knowledge Exchange: http://www.niagaraknowledgeexchange.com/wp-content/uploads/sites/2/2018/07/2018-07-24-Niagara-Counts-2018.pdf
- [Background] Davidson L, Bellamy C, Guy K, Miller R. Peer support among persons with severe mental illnesses: a review of evidence and experience. World Psychiatry. 2012 Jun;11(2):123-8. doi: 10.1016/j.wpsyc.2012.05.009. PMID 22654945
- [Background] de Vet R, van Luijtelaar MJ, Brilleslijper-Kater SN, Vanderplasschen W, Beijersbergen MD, Wolf JR. Effectiveness of case management for homeless persons: a systematic review. Am J Public Health. 2013 Oct;103(10):e13-26. doi: 10.2105/AJPH.2013.301491. Epub 2013 Aug 15. PMID 23947309
- [Background] Dennis ML, Chan YF, Funk RR. Development and validation of the GAIN Short Screener (GSS) for internalizing, externalizing and substance use disorders and crime/violence problems among adolescents and adults. Am J Addict. 2006;15 Suppl 1(Suppl 1):80-91. doi: 10.1080/10550490601006055. PMID 17182423
- [Background] Forchuk C, Reiss JP, Mitchell B, Ewen S, Meier A. Homelessness and housing crises among individuals accessing services within a Canadian emergency department. J Psychiatr Ment Health Nurs. 2015 Aug;22(6):354-9. doi: 10.1111/jpm.12212. Epub 2015 May 20. PMID 25990385
- [Background] Ford I, Norrie J. Pragmatic Trials. N Engl J Med. 2016 Aug 4;375(5):454-63. doi: 10.1056/NEJMra1510059. No abstract available. PMID 27518663
- [Background] Forthofer, R. N., Lee, E. S., & Hernandez, M. (2007). Biostatistics : A Guide to Design, Analysis, and Discovery (Second ed.). Amsterdam: Elsevier Ltd. Retrieved from http://search.ebscohost.com/login.aspx?direct=true&db=nlebk&AN=185748&site=ehost-live
- [Background] Hakanson C, Ohlen J. Illness narratives of people who are homeless. Int J Qual Stud Health Well-being. 2016 Nov 30;11:32924. doi: 10.3402/qhw.v11.32924. eCollection 2016. PMID 27914194
- [Background] Hughes NR. Are institutional health policies exclusionary? Qual Health Res. 2014 Mar;24(3):366-74. doi: 10.1177/1049732314523504. Epub 2014 Feb 18. PMID 24549411
- [Background] Hwang SW, Martin RE, Tolomiczenko GS, Hulchanski JD. The relationship between housing conditions and health status of rooming house residents in Toronto. Can J Public Health. 2003 Nov-Dec;94(6):436-40. doi: 10.1007/BF03405081. PMID 14700243
- [Background] Irestig R, Burstrom K, Wessel M, Lynoe N. How are homeless people treated in the healthcare system and other societal institutions? Study of their experiences and trust. Scand J Public Health. 2010 May;38(3):225-31. doi: 10.1177/1403494809357102. Epub 2010 Jan 7. PMID 20056785
- [Background] Janssen MF, Pickard AS, Golicki D, Gudex C, Niewada M, Scalone L, Swinburn P, Busschbach J. Measurement properties of the EQ-5D-5L compared to the EQ-5D-3L across eight patient groups: a multi-country study. Qual Life Res. 2013 Sep;22(7):1717-27. doi: 10.1007/s11136-012-0322-4. Epub 2012 Nov 25. PMID 23184421
- [Background] Larson CO. Use of the SF-12 instrument for measuring the health of homeless persons. Health Serv Res. 2002 Jun;37(3):733-50. doi: 10.1111/1475-6773.00046. PMID 12132603
- [Background] Lauber C, Lay B, Rossler W. Homeless people at disadvantage in mental health services. Eur Arch Psychiatry Clin Neurosci. 2006 Apr;256(3):138-45. doi: 10.1007/s00406-005-0616-4. PMID 16639520
- [Background] Loudon K, Treweek S, Sullivan F, Donnan P, Thorpe KE, Zwarenstein M. The PRECIS-2 tool: designing trials that are fit for purpose. BMJ. 2015 May 8;350:h2147. doi: 10.1136/bmj.h2147. No abstract available. PMID 25956159
- [Background] Mills ED, Burton CD, Matheson C. Engaging the citizenship of the homeless-a qualitative study of specialist primary care providers. Fam Pract. 2015 Aug;32(4):462-7. doi: 10.1093/fampra/cmv036. Epub 2015 May 22. PMID 26002771
- [Background] Misch DA. Basic strategies of dynamic supportive therapy. J Psychother Pract Res. 2000 Fall;9(4):173-89. PMID 11069130
- [Background] Neumann, P. J., Sanders, G. D., Russell, L. B., Siegel, J. E., & Ganiats, T. G. (2017). Cost-effectiveness in health and medicine (Second ed.). Oxford: Oxford University Press.
- [Background] Niagara Counts. (2018, March 15). Retrieved from https://www.niagararegion.ca/social-services/niagara-counts.aspx
- [Background] Nicholas DB, Newton AS, Calhoun A, Dong K, deJong-Berg MA, Hamilton F, Kilmer C, McLaughlin AM, Shankar J. The Experiences and Perceptions of Street-Involved Youth Regarding Emergency Department Services. Qual Health Res. 2016 May;26(6):851-62. doi: 10.1177/1049732315577605. Epub 2015 Mar 31. PMID 25829466
- [Background] Nickasch B, Marnocha SK. Healthcare experiences of the homeless. J Am Acad Nurse Pract. 2009 Jan;21(1):39-46. doi: 10.1111/j.1745-7599.2008.00371.x. PMID 19125894
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Raven MC, Kushel M, Ko MJ, Penko J, Bindman AB. The Effectiveness of Emergency Department Visit Reduction Programs: A Systematic Review. Ann Emerg Med. 2016 Oct;68(4):467-483.e15. doi: 10.1016/j.annemergmed.2016.04.015. Epub 2016 Jun 8. PMID 27287549
- [Background] Redelmeier DA, Molin JP, Tibshirani RJ. A randomised trial of compassionate care for the homeless in an emergency department. Lancet. 1995 May 6;345(8958):1131-4. doi: 10.1016/s0140-6736(95)90975-3. PMID 7723543
- [Background] Repper J, Carter T. A review of the literature on peer support in mental health services. J Ment Health. 2011 Aug;20(4):392-411. doi: 10.3109/09638237.2011.583947. PMID 21770786
- [Background] Riddell MA, Renwick C, Wolfe R, Colgan S, Dunbar J, Hagger V, Absetz P, Oldenburg B; Australasian Peers for Progress Diabetes Project Investigators. Cluster randomized controlled trial of a peer support program for people with diabetes: study protocol for the Australasian Peers for Progress study. BMC Public Health. 2012 Oct 4;12:843. doi: 10.1186/1471-2458-12-843. PMID 23035666
- [Background] Miller WR, Rollnick S. Ten things that motivational interviewing is not. Behav Cogn Psychother. 2009 Mar;37(2):129-40. doi: 10.1017/S1352465809005128. PMID 19364414
- [Background] Saab D, Nisenbaum R, Dhalla I, Hwang SW. Hospital Readmissions in a Community-based Sample of Homeless Adults: a Matched-cohort Study. J Gen Intern Med. 2016 Sep;31(9):1011-8. doi: 10.1007/s11606-016-3680-8. Epub 2016 May 19. PMID 27197973
- [Background] Shumway M, Boccellari A, O'Brien K, Okin RL. Cost-effectiveness of clinical case management for ED frequent users: results of a randomized trial. Am J Emerg Med. 2008 Feb;26(2):155-64. doi: 10.1016/j.ajem.2007.04.021. PMID 18272094
- [Background] Stergiopoulos V, Gozdzik A, Cohen A, Guimond T, Hwang SW, Kurdyak P, Leszcz M, Wasylenki D. The effect of brief case management on emergency department use of frequent users in mental health: Findings of a randomized controlled trial. PLoS One. 2017 Aug 3;12(8):e0182157. doi: 10.1371/journal.pone.0182157. eCollection 2017. PMID 28771524
- [Background] Sun S, Irestig R, Burstrom B, Beijer U, Burstrom K. Health-related quality of life (EQ-5D) among homeless persons compared to a general population sample in Stockholm County, 2006. Scand J Public Health. 2012 Mar;40(2):115-25. doi: 10.1177/1403494811435493. Epub 2012 Feb 10. PMID 22327187
- [Background] Sunderland, K., Mishkin, W., & Peer Leadership Group. (2013). Guidelines for the Practice and Training of Peer Support. Calgary, AB: Mental Health Commission of Canada. Retrieved from: http://www.mentalhealthcommission.ca
- [Background] Tango, T. (2009). Sample size formula for randomized controlled trials with counts of recurrent events. Statistics & Probability Letters, 79(4), 466-472. doi:10.1016/j.spl.2008.09.016
- [Background] Vingilis E, Hartford K, Diaz K, Mitchell B, Velamoor R, Wedlake M, White D. Process and outcome evaluation of an emergency department intervention for persons with mental health concerns using a population health approach. Adm Policy Ment Health. 2007 Mar;34(2):160-71. doi: 10.1007/s10488-006-0093-8. Epub 2006 Oct 6. PMID 17024576
- [Background] Wen CK, Hudak PL, Hwang SW. Homeless people's perceptions of welcomeness and unwelcomeness in healthcare encounters. J Gen Intern Med. 2007 Jul;22(7):1011-7. doi: 10.1007/s11606-007-0183-7. Epub 2007 Apr 6. PMID 17415619
- [Background] Xie F, Pullenayegum E, Gaebel K, Bansback N, Bryan S, Ohinmaa A, Poissant L, Johnson JA; Canadian EQ-5D-5L Valuation Study Group. A Time Trade-off-derived Value Set of the EQ-5D-5L for Canada. Med Care. 2016 Jan;54(1):98-105. doi: 10.1097/MLR.0000000000000447. PMID 26492214